CLINICAL TRIAL: NCT05359250
Title: Evaluation of Myocardial Dysfunction Due to mRNA-based SARS-CoV-2 Vaccines
Brief Title: Myocardial Injury and Dysfunction Associated With COVID-19 Vaccination
Acronym: MIDAVAX
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Collaborators: American Heart Association (Other); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Other Study IDs: 21-4055; 3UM1AI068614-14S1 (NIH)
Record Dates: First submitted 2022-05-02; First posted 2022-05-03 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Myocardial Injury; COVID-19; Vaccine Reaction
Keywords: COVID-19; mRNA vaccines; myocardial injury; myocarditis; gene expression
MeSH Terms: conditions — COVID-19; Myocarditis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — Right heart catheterization will be performed and a small sample from right ventricle distal septum will be collected. The endomyocardial biopsy sample will be processed for RNA extraction and gene expression.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with evidence of myocardial injury related to vaccination with a SARS-CoV-2 mRNA vaccine: Patients who present with new symptoms of chest pain within 2-10 days following SARS-CoV-2 mRNA vaccination will be recruited up to 180 days following diagnosis. Patients will be screened using multiple methods and then provided informed consent. If patients are unable to consent, health care decision makers of patients who meet initial inclusion criteria will be approached for consent. Following informed consent, a cardiac MRI will be performed (if not performed prior) to assess myocardial function and potential damage. Patients will qualify on the basis of the presence of late-gadolinium enhancement and/or abnormal T1 mapping on MRI. The patient will then be taken to the cardiac catheterization lab where he/she will undergo endomyocardial biopsy and right heart catheterization (RHC) for candidate gene analysis. A blood sample will be collected to analyze circulating biomarkers associated with myocardial injury.

SUMMARY:
The overall goal of the study is to investigate the characteristics and potential mechanisms responsible for myocardial injury and dysfunction in patients after COVID-19 vaccination. Cardiac damage will be assessed with cardiac MRI and endomyocardial biopsy (EmBx) histopathology. Myocardial gene expression will be measured in RNA extracted from EmBxs mRNA abundance compared to nonfailing and failing control hearts.

DETAILED DESCRIPTION:
To determine whether there is microvascular thrombosis-associated myocardial damage and dysfunction vs. inflammation or other changes in patients who, following administration of SARS-CoV-2 mRNA vaccine, develop evidence of myocardial injury typically diagnosed as "myocarditis" based on cardiac MRI findings.

Further, the degree of inflammatory reaction vs. microthrombotic injury to cardiac myocytes from biopsied myocardial tissue will be compared with biopsied myocardial tissue from control hearts. mRNA expression of the ACE2 and ITGA5 binding targets of SARS-Cov-2 Spike protein encoded by mRNA vaccines, as well as expression of other genes that may contribute to post-vaccine pro-thrombotic and pro-inflammatory states including Coagulation Factor 3 (F3, also known as tissue factor), ACE, AGTR1 and AGT) or a dysfunctional cardiac state (NPPB as a marker of pathologic remodeling) will be examined as candidate genes. Additional, global gene expression is being measured by RNA-Seq and microarray.

ELIGIBILITY:
Inclusion Criteria:

1. age ≥18 years;
2. clear evidence of myocardial involvement including:

   1. High Sensitivity Troponin I value of (≥0.05 ng/ml (the 99% upper bound)) OR
   2. an LVEF < 50% OR
   3. ST-T change suggesting STEMI, NSTEMI or myopericarditis in the absence of coronary artery disease, OR
   4. new onset sustained VT or VF
3. Late gadolinium enhancement or edema on cMRI consistent with myocardial injury or inflammation.
4. Documentation of vaccination with mRNA-based COVID-19 vaccine.
5. No history of COVID-19, or a negative SARS-CoV-2 PCR or other FDA approved laboratory test within 1 week of enrollment.
6. Patient and/or legally authorized representative must be competent to understand and agree with informed consent form.

Exclusion Criteria:

1. Hemodynamic instability as evidenced by escalating doses of inotropic agents or vasopressors within the prior 24 hours
2. Respiratory instability as evidenced by increasing oxygen requirements over the 24 hours prior to consent or FiO2 requirement ≥ 60 %.
3. evidence that respiratory failure is the primary reason for myocardial dysfunction;
4. Moderate to severe pulmonary hypertension (mean PAP ≥35 mmHg);
5. INR >1.8 on no anticoagulation or contraindication to withdrawing anticoagulation;
6. platelets <100,000/mm3.
7. History of laboratory-confirmed SARS-CoV-2 infection as determined by polymerase chain reaction (PCR) testing or other commercial or public health assay.
8. Acute or chronic kidney disease with glomerular filtration rate < 30 ml/min.1.72m2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Ten patients with new symptoms of chest discomfort and biomarkers of myocardial injury that occurred 2-10 days following SARS-CoV-2 mRNA vaccination will be recruited up to 180 days following diagnosis. Patients will have no other known etiology for myocardial injury other than recent mRNA COVID vaccine exposure. Patients may be referred from inpatient or outpatient settings, from across the UCHealth system, but will be recruited in-person at University of Colorado Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2021-05-12 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Myocardial damage | clinical follow up for at least 30 days following endomyocardial biopsy
  Initial clinical diagnosis of myocardial injury or myocarditis will be confirmed by cardiac MRI. Specific findings of late gadolinium enhancement and abnormal T1-signals within the myocardium consistent with acute injury, inflammation or edema will be evaluated.
Histopathological changes assessed by light- and electron-microscopy in myocardial tissue | clinical follow up for at least 30 days following endomyocardial biopsy
  Determining the histopathologic changes present in the endomyocardial biopsies of patients with COVID-19 vaccine-induced myocardial injury. Assessment of the standard H&E stains will include evaluation for presence and degree of inflammation within the myocardium, presence of microvascular thrombi within vasculature, and evidence of myocardial damage. The trichrome, iron, and Congo red stains will be used to evaluate for the presence of fibrosis, iron, or amyloid, respectively. Electron microscopy will be employed to examine cardiac myocyte and small blood vessel architectures.
Myocardial mRNA expression | clinical follow up for at least 30 days following endomyocardial biopsy
  Measure myocardial mRNA expression of candidate genes involved in Spike protein binding and cell entry (ACE2 and ITGA5), the renin-angiotensin system (ACE, AGT, AGTR1), initiation of coagulation (F3/TF) and pathologic myocardial remodeling (NPPB).

SECONDARY OUTCOMES:
Myocardial mRNA expression of additional genes measured by both RNA-Seq and microarray. | clinical follow up for at least 30 days following endomyocardial biopsy
  Measure mRNA expression of additional candidate and global genes, and compare results to nonfailing and failing controls. Seven candidate genes will be measured by three platforms (qPCR, RNA-Seq and microarray), and global transcripts by RNA-Seq and microarray.

CONTACTS AND LOCATIONS:
Overall Officials: Natasha Altman, MD, Principal Investigator — University of Colorado, Denver; Bristow Michael, MD/PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Anschutz Medical Campus, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Patone M, Mei XW, Handunnetthi L, Dixon S, Zaccardi F, Shankar-Hari M, Watkinson P, Khunti K, Harnden A, Coupland CAC, Channon KM, Mills NL, Sheikh A, Hippisley-Cox J. Risks of myocarditis, pericarditis, and cardiac arrhythmias associated with COVID-19 vaccination or SARS-CoV-2 infection. Nat Med. 2022 Feb;28(2):410-422. doi: 10.1038/s41591-021-01630-0. Epub 2021 Dec 14. PMID 34907393
- [Background] Oster ME, Shay DK, Su JR, Gee J, Creech CB, Broder KR, Edwards K, Soslow JH, Dendy JM, Schlaudecker E, Lang SM, Barnett ED, Ruberg FL, Smith MJ, Campbell MJ, Lopes RD, Sperling LS, Baumblatt JA, Thompson DL, Marquez PL, Strid P, Woo J, Pugsley R, Reagan-Steiner S, DeStefano F, Shimabukuro TT. Myocarditis Cases Reported After mRNA-Based COVID-19 Vaccination in the US From December 2020 to August 2021. JAMA. 2022 Jan 25;327(4):331-340. doi: 10.1001/jama.2021.24110. PMID 35076665